CLINICAL TRIAL: NCT04523610
Title: Telehealth Intervention Program for Older Adults (TIP-OA) Struggling With Mental Health/Cognitive Issues
Brief Title: Telehealth Intervention Program for Older Adults
Acronym: TIP-OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Soham Rej MD, MSc, Principal Investigator, Lady Davis Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TIP-OA
Record Dates: First submitted 2020-07-16; First posted 2020-08-21 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2020-09

CONDITIONS: Depression, Anxiety; Cognitive Impairment; Stress
Keywords: Mental Health; Teleheath; Volunteer; COVID-19; Older Adults
MeSH Terms: conditions — Depression; Anxiety Disorders; Cognitive Dysfunction; Psychological Well-Being; COVID-19

STUDY DESIGN:
Intervention Model Description: This is a mixed-methods (qualitative and quantitative) model
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Program Users - Quantitative (Experimental): The Telehealth Intervention Program (TIP-OA) for older adults was created during the COVID-19 pandemic to support the health of older adults who are isolated or have mental health/cognitive issues. Within the TIP-OA program, trained volunteers provide friendly phone calls once a week to older adults (age 60+). 200 participants will be recruited for the quantitative component of the study.
  Interventions: Behavioral: Telehealth phone calls
- Program Users - Qualitative (Other): Interviews will be conducted with 25 participants regarding their perceptions and experiences in the TIP-OA program.
  Interventions: Behavioral: Telehealth phone calls
- Volunteers - Qualitative (Other): 15 volunteers taking part in the semi-structured interviews and 16 volunteers participating in the focus groups. The interviews and focus groups will evaluate their roles, experiences, and challenges volunteering with the TIP-OA program.
  Interventions: Other: Volunteer of TIP-OA Program
- Stakeholders - Qualitative (Other): 18 stakeholders (clinicians, community partners, TIP-OA team members) will participate in focus groups and interviews. Specifically, 10 clinicians will participate in one focus group and 8 community partners/team members will participate in interviews. The interviews and focus groups will evaluate their roles, experiences, and challenges volunteering with the TIP-OA program.
  Interventions: Other: Stakeholder of TIP-OA Program

INTERVENTIONS:
Behavioral: Telehealth phone calls — The volunteer-based weekly Telehealth support primarily provides program users with friendly listening/conversation. Volunteers will also inquire about their general wellbeing, provide information about COVID-19, and ask if the older adult needs any help or support (e.g. food delivery, medication from their pharmacy).
  Arms: Program Users - Qualitative; Program Users - Quantitative
Other: Volunteer of TIP-OA Program — Participant is a volunteer of the TIP-OA Program
  Arms: Volunteers - Qualitative
Other: Stakeholder of TIP-OA Program — Participant is a stakeholder of the TIP-OA Program
  Arms: Stakeholders - Qualitative

SUMMARY:
COVID-19 is having profound effects on older adults' due to social isolation measures which may negatively impact individuals' mental and physical health. Recently, a telephone program, the Telehealth Intervention Program for Older Adults (TIP-OA), was created. In this program, a volunteer is calling older adults (age≥60) every week to have a friendly conversation. The objective of this study is to evaluate the effectiveness of this telephone program (TIP-OA) in reducing stress, improving the mental health of program users, and understand their experiences.

DETAILED DESCRIPTION:
Social isolation has profound negative impacts on the mental health of older adults (generally those aged ≥60), such as stress, anxiety, cognitive decline, and depression. Depression is the #1 cause of disability worldwide. Prior to the pandemic, mental disorders were affecting >10-15% older adults and more than 1,000,000 Canadians, with an estimated annual cost of $15 billion, which will increase with COVID-19.

There are 4.5 billion people globally in voluntary confinement and practicing social distancing. Older adults are more isolated and face risks to their health: i.e. increased risk for depression, ER visits and hospital admissions. Older isolated individuals are 4-5 times more likely to be rehospitalized. Moreover, older adults with stress, anxiety, and/or depression, have 50% higher healthcare costs and at 2 times increased mortality. Together these factors threaten to further overwhelm a healthcare system already strained from managing the direct morbidity and mortality of COVID-19.

During the pandemic, with an increased burden on health professionals who can be burnt out, reassigned, or infected with COVID-19, engaging lay volunteers may be beneficial to increase capacity. During COVID, many people are currently unable to work/study, are underemployed/unemployed, and able to volunteer. In a low-resource part of India, an in-person lay volunteer intervention was able to improve depression and other mental health symptoms in older adults. However, a systematic review of volunteer interventions in older individuals with mental health found that the evidence-base is limited with small sample sizes, few randomized controlled trials, especially for remote service delivery. Telehealth has been successful in connecting with socially isolated adults. Telehealth can be adopted in areas where healthcare access is limited and has evidence for improving depression and anxiety. However, telehealth programs that use the internet, tablets, smartphones apps or computers may not be accessible to or preferred by older adults; a survey of 500 older adults found that while only 10% used the internet, 77% did own a mobile phone. In the current COVID-19 context, many such interventions are not feasible for rapid implementation due to lack of infrastructure, training, and low rates of digital literacy in older adults. In a telephoning initiative prior to COVID, older isolated adults reported forming satisfying relationships as well as gaining confidence, engaging in the community and being more socially active. Given these limitations and need for immediate support for vulnerable older adults facing isolation during COVID-19, telephone-based support with volunteers is considered a potential fast, inexpensive, scalable, and convenient intervention option requiring further investigation.

The Telehealth Intervention Program (TIP-OA) for older adults was created during the COVID-19 pandemic to support the health of older adults who are isolated or have mental health/cognitive issues. Within the TIP-OA program, volunteers provide friendly phone calls once a week to older adults (age 60+).

The TIP-OA program provides once a week friendly phone calls from trained volunteers to older adults (age 60+), particularly to older adults struggling with mental health/cognitive issues. The clinical program does not provide any kind of treatment to the program user. Rather, the volunteer-based friendly telephone/telehealth calls adopt a simple and proactive communication technique: e.g., calling seniors to inquire about their general wellbeing, giving out information about COVID-19, asking if the seniors need any help or support (e.g. food delivery, medication from their pharmacy), connecting seniors with community organizations offering services (e.g. grocery delivery), or just talking and giving friendly company on the phone to increase a sense of connection. Moreover, program users are given a phone number for queries, comments, or complaints regarding the program or their volunteer. This study evaluates the effectiveness of the clinical service TIP-OA in 1) reducing stress (Perceived Stress Scale), 2) improving the mental health of service users (Patient Health Questionnaire-9, Generalized Anxiety Disorder-7, Fear of COVID-19 Scale), 3) improving mental healthcare utilization (e.g. hospital visits, hospitalizations, and outpatient visits), 4) compare mental health outcomes based on service users baseline risk, as well as 5) understand the experiences of service users, volunteers, and other stakeholders to improve TIP-OA and related future programs.

Using mixed-methods, the impact of the program will be evaluated systematically. The investigators will assess mental health outcomes in 200 older adults at baseline, 4- and 8-weeks (primary study endpoint). In addition, the investigators will perform qualitative analyses focus groups and/or individual semi-structured interviews with older adult participants, volunteers, community partners, and team members. The investigators anticipate that the TIP-OA program will be associated with improvements in stress, anxiety, and depression. If this is indeed the case, the investigators hope to share results with colleagues who could also develop similar programs internationally.

ELIGIBILITY:
Inclusion Criteria: Program Users

* TIP-OA Program User
* Aged ≥60 years
* Residing in Montreal
* Speak English or French
* Capable of giving consent (judged by a member of the research team to adequately understand information relevant in making a decision about research participation, and to reasonably appreciate foreseeable consequences of a decision or lack of decision)

Exclusion Criteria: Program Users

* Not capable of giving consent (vetted for this by the clinician team)

Inclusion Criteria: Volunteers

* TIP-OA program volunteer
* Able to speak English or French

Exclusion Criteria: Volunteers

* None

Inclusion Criteria: Stakeholders

* TIP-OA program stakeholder (community partners, program organizers, and clinicians)
* Able to speak English or French

Exclusion Criteria: Stakeholders

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | Change from Baseline to 4- and 8-weeks (15 minute assessment)
  Perceived Stress Scale (PSS) is a 14-item scale used to measure the degree to which life events are experienced and appraised as stressful. It asks respondents about how often they have felt certain ways in the past month, with responses ranging from 0 (never) to 4 (very often).
Patient Health Questionnaire-9 (PHQ-9) | Change from Baseline to 4- and 8-weeks (15 minute assessment)
  Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report questionnaire used to diagnose depression and assess symptom severity. The questionnaire asks individuals how often in the last two weeks they have been bothered by problems like "feeling down, depressed, and hopeless" and "poor appetite or overeating." Scores for each question include 0 (not at all), 1 (several days), 2 (more than half of the days), and 3 (nearly every day).
Generalized Anxiety Disorder-7 (GAD-7) | Change from Baseline to 4- and 8-weeks (15 minute assessment)
  Generalized Anxiety Disorder-7 (GAD-7) is a 7-item scale that measures symptoms of anxiety present in the previous 2 weeks. Respondents can choose from a score of 0 (not at all sure), 1 (several days), 2 (over half the days), or 3 (nearly every day). Items include "Not being able to stop or control worrying" and "Being so restless that it's hard to sit still".
Fear of COVID-19 Scale | Change from Baseline to 4- and 8-weeks (15 minute assessment)
  Fear of COVID-19 Scale is an 18-item scale measuring individuals' anxiety, fear and concern surrounding the COVID-19 pandemic. Items include: "Fear that I will be infected" and "Worry if I will be assigned to COVID wards if hospitalized" (34).
Mental Healthcare Utilization | Assessed in the 8 weeks prior to baseline and during the 8-week follow-up
  Mental healthcare utilization will be assessed using medical records, including the number of ER visits, hospitalizations, and outpatient visits

SECONDARY OUTCOMES:
Interviews and Focus Groups with Volunteers | 8-weeks (2 hours)
  What are the roles, contributions, and challenges of volunteers in identifying the needs of program users and volunteers, providing access to services, and creating appropriate responses to identified needs for the success and efficacy of the program?
Interviews and Focus Groups with Stakeholders | 8-weeks (2 hours)
  What are the roles, contributions, and challenges of different stakeholders (e.g. community partners, program organizers, and clinicians) in identifying the needs of program users and volunteers, providing access to services, and creating appropriate responses to identified needs for the success and efficacy of the program?
Interviews with Program Users | 8-weeks (2 hours)
  What are the experiences and evaluation of the program users about their engagement with the TIP-OA? Has the program contributed in improving the health of the program users?

CONTACTS AND LOCATIONS:
Overall Officials: Soham Rej, MD/MSc, Principal Investigator — Lady Davis Institute
Locations (1):
- Institute of Community and Family Psychiatry, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dikaios E, Sekhon H, Allard A, Vacaflor B, Goodman A, Dwyer E, Lavin-Gonzalez P, Mahdanian A, Park H, Walsh C, Sasi N, Nazar R, Gruber J, Su CL, Hanganu C, Royal I, Schiavetto A, Cinalioglu K, Rigas C, Launay C, Beauchet O, McDonald E, Seitz D, Kumar S, Nair V, Miresco M, Bruneau MA, Alexopoulos G, Looper K, Vahia I, Rej S, Bukhari SN. Connecting During COVID-19: A Protocol of a Volunteer-Based Telehealth Program for Supporting Older Adults' Health. Front Psychiatry. 2020 Dec 2;11:598356. doi: 10.3389/fpsyt.2020.598356. eCollection 2020. PMID 33343425